CLINICAL TRIAL: NCT01309230
Title: Open-label Phase II Trial of Adjuvant bishRNAfurin and GMCSF Augmented Autologous Tumor Cell Vaccine (FANG™) for High Risk Stage III/IV Ovarian Cancer
Brief Title: A Trial of FANG™ Vaccine for Participants With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL 105
Record Dates: First submitted 2011-02-25; First posted 2011-03-07 (Estimated); Results first posted 2023-03-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer
Keywords: Stage III; Stage IV; epithelial ovarian cancer; ovarian cancer; Adjuvant bi-shRNAfurin and GMCSF; immunotherapy; Vigil; FANG; Autologous Tumor Cell Vaccine
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — FANG vaccine

STUDY DESIGN:
Intervention Model Description: Participants were randomized 2 (Group A (Vigil)):1 (Group B (Standard of Care)). Randomization was only applicable to participants enrolled prior to approval of Protocol Amendment 8, dated June 19, 2014. All participants enrolled after approval of Protocol Amendment 8 were assigned to Group A (Vigil).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Vigil™) (Experimental): Vigil immunotherapy was administered at a concentration of at 1 x 10e7 cells/injection via intradermal injection for a minimum of 4 doses and a maximum of 12 doses starting ≥3 weeks following completion of chemotherapy (no longer than 2.5 months post chemotherapy). Participants were treated monthly for up to 12 months as long as sufficient Vigil was available and the participant was clinically stable.
  Interventions: Biological: Vigil™
- Group B (Observational - Standard of Care) (No Intervention): Participants received standard of care without maintenance therapy.

INTERVENTIONS:
Biological: Vigil™ — Vigil is composed of autologous tumor cells harvested from the patient at the time of initial de-bulking surgery which are then transfected extracorporeally, with a plasmid encoding for the gene for GM-CSF, an immune-stimulatory cytokine, and a bifunctional, short hairpin RNA which specifically knocks down the expression of furin, the critical convertase responsible for production of the two TGβ isoforms.
  Other Names: formerly known as FANG™ vaccine; Bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Immunotherapy
  Arms: Group A (Vigil™)

SUMMARY:
This was a clinical trial for women with ovarian cancer scheduled to have an operation to remove the cancerous tissue. The cancer cells removed during the planned surgery were used to attempt to make the investigational product, named Vigil. Vigil is considered an immunotherapy. In this study, participants who met the requirements to be in the study and if Vigil was successfully made from the participants cancer cells, participants underwent treatment with their standard chemotherapy regimen. At the end of the standard chemotherapy regimen and if there was no evidence of remaining cancer, participants were randomly assigned to receive the Vigil or would be assigned to the standard of care group, which in this study meant no further treatment was given to the participant.

The purpose of this study was to compare the difference between the participants who received Vigil versus the usual care after completion of standard chemotherapy and to determine if Vigil delayed or prevented ovarian cancer from coming back.

DETAILED DESCRIPTION:
This was a Phase II open-label study of Vigil™ autologous tumor cell vaccine trial administered to women with Stage III/IV epithelial ovarian cancer. Tumor was harvested at the time of surgical debulking (standard of medical care). Participants who achieved clinical complete response (CR) following primary surgical debulking and front-line doublet chemotherapy were randomized 2:1 to either treatment with Vigil (Group A) or standard of care without maintenance therapy (Group B). After randomization, participants were stratified into cohorts by baseline CA-125 (greater than 10 to less than 20 units/mL versus less than or equal to 10 units/mL). For data analysis, participants could further be stratified by surgical stage (Stage IV or suboptimal debulking (> 1cm residual), Stage III disease versus Stage III disease with optimal debulking (< 1cm residual). Participants enrolled in Group A (Vigil) received 1.0 x 10e7 cells / intradermal injection of gene transfected autologous tumor cells, Vigil™, once a month for up to 12 doses as long as sufficient material was available or until trial endpoints were met. Enough harvested tissue to provide a minimum of 4 monthly injections was required for entry into the study. Participants enrolled in Group B (Standard of Care, SOC) were observed and assessed until trial endpoints were met. Protocol Amendment 8, June 19, 2014 removed randomization such that all patients screening for enrollment into the main portion of the trial (including those who previously had tumor tissue harvested) would be assigned to Group A (Vigil).

Both groups of participants were seen once a month in an outpatient setting. Hematologic function, liver enzymes, renal function and electrolytes were monitored monthly. Immune function analysis including ELISPOT analysis of cytotoxic T cell function to autologous tumor antigens were monitored at (≤ 24 hours before the third cycle chemotherapy (post debulking), baseline (screening); prior to Vigil injection at Months 2, 3, 6 and EOT. CA-125 was monitored at baseline, every month for the first year, every 3 months +/- 2 weeks for the second and third year.

Participants assigned to group A were allowed to continue treatment with Vigil until disease recurrence or exhaustion of the patient's vaccine supply. If ≥ Grade 2 toxicity by NCI Common Toxicity Criteria (excluding Grade 2 fever ≤ 24 hours and Grade 2 and 3 injection site reactions) developed related to study treatment, the vaccine dose was reduced by 50% and continued on a monthly basis.

Efficacy assessments included time to disease recurrence, immune surrogate markers, and quality of life questionnaire (FACT-O, Version 4). Safety assessments included physical examination, performance status, and vital signs. Adverse events were recorded using CTCAE version 3.

ELIGIBILITY:
Tissue Inclusion Criteria

Patients were eligible for tissue procurement for the Vigil™ vaccine manufacturing process if they met all of the following criteria:

1. Presumptive Stage III/IV papillary serous or endometrioid ovarian cancer.
2. Per Amendment #8, treatment naïve, high risk ovarian cancer was no longer be stratified, but the following information was collected:

   1. Stage IV or suboptimal (>1 cm residual) Stage III disease versus Stage III patients with optimal (≤1 cm residual) disease,
   2. CA-125 ≤10 U/ml versus CA-125 greater than 10 but less than or equal to 20 U/ml
   3. IP chemotherapy versus IV chemotherapy
3. Availability of "golf-ball" size 10-30 grams tissue at time of primary surgical debulking.
4. ECOG performance status (PS) 0-2 prior to tumor debulking laparotomy
5. Ability to understand and the willingness to sign a written informed consent document for tissue harvest.

Tissue Exclusion Criteria

Patients who met any of the following criteria were not eligible for tissue procurement for the Vigil manufacturing:

1. Medical condition requiring any form of chronic systemic immunosuppressive therapy (steroid or other) except physiologic replacement doses of hydrocortisone or equivalent (no more than 30 mg hydrocortisone or 10 mg prednisone equivalent daily) for < 30 days duration.
2. Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers were allowed if definitively resected.
3. Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 2 months.
4. Any documented history of autoimmune disease with exception of Type 1 diabetes on stable insulin regimen, hypothyroidism on stable dose of replacement thyroid medication, vitiligo, or asthma not requiring systemic steroids.
5. Known HIV or chronic Hepatitis B or C infection.
6. Known history of allergies or sensitivities to gentamicin.
7. History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or was not in the best interest of the patient to participate, in the opinion of the treating Investigator.

Study Enrollment Inclusion Criteria

Patients were registered for inclusion in this study if they met all of the following criteria:

1. Histologically confirmed Stage III/IV papillary serous or endometrioid ovarian cancer.
2. Clinically defined CR (no cancer related symptoms, normal physical examination and CT scan abdomen/pelvis and CXR, and CA-125 ≤20 U/ml) following completion of primary surgical debulking. Patients enrolled must have completed at least 5 but no more than 6 cycles platinum/taxane adjuvant or interval debulking and chemotherapy (or chemotherapy as per recommendations of NCCN guidelines, category 1 (IP chemotherapy included)). (Patients who completed surgery/chemotherapy with a CA-125 >20 U/mL pre-registration had the option of being followed up to 2 months if serial CA-125 values continued to decrease at a rate of CA-125 decrease of ≥ 50% per month.)
3. Successful manufacturing of 4 vials of Vigil™ vaccine
4. Recovered from all clinically relevant toxicities related to prior protocol specific therapies (including neuropathy to ≤Grade 2).
5. ECOG performance status (PS) 0-1.
6. Normal organ and marrow function as defined below:

   Absolute granulocyte count ≥ 1,500/mm3 Absolute lymphocyte count ≥ 200/mm3 Platelets ≥ 75,000/mm3 Total bilirubin ≤ 2 mg/dL AST(SGOT)/ALT(SGPT) ≤ 2x institutional upper limit of normal Creatinine < 1.5 mg/dL
7. Patients must have been off all "statin" drugs for ≥ 2 weeks prior to initiation of therapy.
8. Ability to understand and the willingness to sign a written informed protocol specific consent document.

Study Enrollment Exclusion Criteria

Patients were excluded from this study if they met any of the following criteria:

1. Surgery involving general anesthesia, radiotherapy, or immunotherapy within 4 weeks prior to randomization. Chemotherapy within 3 weeks prior to Vigil™ vaccine administration. Steroid therapy within 1 week prior to vaccine administration
2. Patients must not have received any other investigational agents within 4 weeks prior to Vigil™ vaccine administration.
3. Patients with history of brain metastases.
4. Patients with compromised pulmonary disease.
5. Short term (<30 days) concurrent systemic steroids ≤ 0.25 mg/kg prednisone per day (maximum 7.5 mg/day) and bronchodilators (inhaled steroids) were permitted; patients requiring other steroid regimens and/or immunosuppressives at randomization were excluded.
6. Prior splenectomy.
7. Prior malignancy (excluding nonmelanoma carcinomas of the skin and carcinoma in situ cervix) unless in remission for ≥ 2 years.
8. Kaposi's Sarcoma.
9. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would have limited compliance with study requirements.
10. Patients with known HIV.
11. Patients with chronic Hepatitis B and C infection.
12. Patients with uncontrolled autoimmune diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-03-08 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Study Director — Gradalis, Inc.
Locations (7):
- United States (7):
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Dartmouth-Hitchcock Medical Center/Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - Texas Oncology - Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Cancer Care Northwest, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Background] Nemunaitis J, Barve M, Orr D, Kuhn J, Magee M, Lamont J, Bedell C, Wallraven G, Pappen BO, Roth A, Horvath S, Nemunaitis D, Kumar P, Maples PB, Senzer N. Summary of bi-shRNA/GM-CSF augmented autologous tumor cell immunotherapy (FANG) in advanced cancer of the liver. Oncology. 2014;87(1):21-9. doi: 10.1159/000360993. Epub 2014 Jun 25. PMID 24968881
- [Background] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Background] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459
- [Background] Ghisoli M, Rutledge M, Stephens PJ, Mennel R, Barve M, Manley M, Oliai BR, Murphy KM, Manning L, Gutierrez B, Rangadass P, Walker A, Wang Z, Rao D, Adams N, Wallraven G, Senzer N, Nemunaitis J. Case Report: Immune-mediated Complete Response in a Patient With Recurrent Advanced Ewing Sarcoma (EWS) After Vigil Immunotherapy. J Pediatr Hematol Oncol. 2017 May;39(4):e183-e186. doi: 10.1097/MPH.0000000000000822. PMID 28338569
- [Background] Rocconi RP, Grosen EA, Ghamande SA, Chan JK, Barve MA, Oh J, Tewari D, Morris PC, Stevens EE, Bottsford-Miller JN, Tang M, Aaron P, Stanbery L, Horvath S, Wallraven G, Bognar E, Manning L, Nemunaitis J, Shanahan D, Slomovitz BM, Herzog TJ, Monk BJ, Coleman RL. Gemogenovatucel-T (Vigil) immunotherapy as maintenance in frontline stage III/IV ovarian cancer (VITAL): a randomised, double-blind, placebo-controlled, phase 2b trial. Lancet Oncol. 2020 Dec;21(12):1661-1672. doi: 10.1016/S1470-2045(20)30533-7. PMID 33271095
- [Result] Oh J, Barve M, Matthews CM, Koon EC, Heffernan TP, Fine B, Grosen E, Bergman MK, Fleming EL, DeMars LR, West L, Spitz DL, Goodman H, Hancock KC, Wallraven G, Kumar P, Bognar E, Manning L, Pappen BO, Adams N, Senzer N, Nemunaitis J. Phase II study of Vigil(R) DNA engineered immunotherapy as maintenance in advanced stage ovarian cancer. Gynecol Oncol. 2016 Dec;143(3):504-510. doi: 10.1016/j.ygyno.2016.09.018. Epub 2016 Sep 24. PMID 27678295
- [Result] Oh J, Barve M, Senzer N, Aaron P, Manning L, Wallraven G, Bognar E, Stanbery L, Horvath S, Manley M, Nemunaitis J, Walter A, Rocconi RP. Long-term follow-up of Phase 2A trial results involving advanced ovarian cancer patients treated with Vigil(R) in frontline maintenance. Gynecol Oncol Rep. 2020 Sep 17;34:100648. doi: 10.1016/j.gore.2020.100648. eCollection 2020 Nov. No abstract available. PMID 33364285
- [Result] Rocconi RP, Stanbery L, Madeira da Silva L, Barrington RA, Aaron P, Manning L, Horvath S, Wallraven G, Bognar E, Walter A, Nemunaitis J. Long-Term Follow-Up of Gemogenovatucel-T (Vigil) Survival and Molecular Signals of Immune Response in Recurrent Ovarian Cancer. Vaccines (Basel). 2021 Aug 12;9(8):894. doi: 10.3390/vaccines9080894. PMID 34452019

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-nine (39) subjects had product manufactured and consented to randomize on CL-PTL-105.
Groups:
- Group A: Vigil™ Alone: Vigil immunotherapy was administered at a concentration of at 1 x 10e7 cells/injection via intradermal injection for a minimum of 4 doses and a maximum of 12 doses starting ≥3 weeks following completion of chemotherapy (no longer than 2.5 months post chemotherapy). Participants were treated monthly for up to 12 months as long as sufficient Vigil was available and the participant was clinically stable.
- Group B: Standard of Care: Participants received standard of care without maintenance therapy.
Period: Overall Study
Arm/Group | Group A: Vigil™ Alone | Group B: Standard of Care
Started | 28 | 11
Completed | 28 | 7
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Observation arm closed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Vigil™) | Group B (Observational - Standard of Care) | Total
Number analyzed (Participants) | 28 | 11 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 7 | 25
  >=65 years | 10 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 11 | 39
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 27 | 11 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 11 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 11 | 39
CA-125 Level [Count of Participants; unit: Participants] — One subject CA-125 value was greater than 20 U/mL, which was outside the inclusion criteria range 0 to 20 U/mL. An exception was granted to allow the subject to enroll as the subject's CA-125 value was below the institutional upper limit of normal which is 34 U/mL.
  Participants
    CA-125 > 10 U/ML but ≤ 20 U/mL | 10 | 8 | 18
    CA-125 ≤ to 10 U/mL | 17 | 3 | 20
    CA-125 > 20 U/mL | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence (TTR)
Description: Time to recurrence is the time to progression by Radiological Tumor Assessment by local investigators using the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1. Disease recurrence was defined as the appearance of any measurable or evaluable lesion or as asymptomatic CA-125 levels >35 U/mL at two consecutive measurements, at least one month apart.
Time Frame: Treatment start to the date of first recurrence or date of death if the participant died before recurrence. Radiographic assessment at baseline, </= 1 week prior to Cycle 4, at Standard of Care intervals, and when CA-125>35 U/mL, approximately 3 years.
Population: Participants who achieved complete clinical response (cCR) at the time of study entry were included in the analysis. After randomization, two participants from Group A were deemed unevaluable as they did not achieve cCR.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Group A (Vigil™): Vigil immunotherapy was administered at a concentration of at 1 x 10e7 cells/injection via intradermal injection for a minimum of 4 doses and a maximum of 12 doses starting ≥3 weeks following completion of chemotherapy (no longer than 2.5 months post chemotherapy). Subjects were treated monthly for up to 12 months as long as sufficient Vigil was available and the subject was clinically stable.
- Group B (Observational - Standard of Care): Subjects received standard of care without maintenance therapy.
Arm/Group | Group A (Vigil™) | Group B (Observational - Standard of Care)
Number analyzed (Participants) | 26 | 11
months | 18.2 [14.7 to 43.4] | 12.4 [10.2 to NA] — N/A = Not Available. Upper confidence interval could not be calculated as there were insufficient number of participants with events.

2. Secondary Outcome: Number of Participants Positive for T-cell and Immune Activation Markers
Description: Gamma interferon (γ-IFN) secretion measured by ELISpot assay was used as a marker for T-cell and immune activation to cancer specific neoantigens. Any participant that had greater than or equal to 10 spots were considered positive.
Time Frame: Blood was collected at tissue procurement, prior to the 1st and 3rd cycles of chemotherapy post debulking, at screening, months 2, 4, 6, end of treatment, and quarterly until recurrence, up to 3 years.
Population: Only participants that were deemed evaluable were included in the analysis. Any participants that were determined to not be in complete response (cCR) after study entry were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Vigil™) | Group B (Observational - Standard of Care)
Number analyzed (Participants) | 26 | 10
Participants | 26 | 0

3. Secondary Outcome: Predictive Potential of Tumor Infiltrating Lymphocyte (TIL) and Tumor Associated Macrophage (TAM) Phenotypes
Description: Predictive potential for TIL and TAM was expected to be measured from tissue collected at baseline and at recurrence.
Time Frame: From tissue procurement until recurrence.
Population: Biopsies were not collected at recurrence, therefore the outcome could not be analyzed. Data were not analyzed.
Arm/Group | Group A (Vigil™) | Group B (Observational - Standard of Care)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Vigil Related Adverse Events (AEs)
Description: AEs were reported using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: From first dose of Vigil until 30 days following last dose of Vigil, up to 13 months.
Population: Participants were counted at most once per preferred term and at most once per system organ class.
Measure: Number; unit: adverse events
Arm/Group | Group A (Vigil™) | Group B (Observational - Standard of Care)
Number analyzed (Participants) | 28 | 11
adverse events
  Grade 3 or higher | 0 | 0
  Grade 2 | 1 | 3
  Grade 1 | 24 | 28

ADVERSE EVENTS:
Time Frame: SAEs and Other Adverse Events: Adverse events were recorded from time of first dose of Vigil (Group A) or from first monthly visit (Group B) and up to 30 days following the last dose study treatment (Group A) or last visit date, up to 13 months. All-cause Mortality: from time of first dose of Vigil and until protocol termination, up to 10 years.
Groups:
- Group A (Vigil™): Participants received Vigil at 1 x 10e7 cells/injection via intradermal injection for a minimum of 4 doses and a maximum of 12 doses. Participants were treated monthly for up to 12 months as long as sufficient Vigil was available and the participant was clinically stable.
Arm/Group | Group A (Vigil™) | Group B (Observational - Standard of Care)
All-Cause Mortality (participants affected / at risk) | 20/28 | 7/11
Serious Adverse Events (participants affected / at risk) | 3/28 | 0/11
Other Adverse Events (participants affected / at risk) | 28/28 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Vigil™) (N=28) | Group B (Observational - Standard of Care) (N=11)
Opiate withdrawal symptoms (General disorders) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Vigil™) (N=28) | Group B (Observational - Standard of Care) (N=11)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Lymphadenopathy cervical (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Ear wax (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic membrane scarring (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyroid nodule (Endocrine disorders) | 1 (1) | 0 (0)
Astigmatism (Eye disorders) | 1 (1) | 0 (0)
Night blindness (Eye disorders) | 1 (1) | 0 (0)
Abdominal bloating (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 4 (5)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Canker sores oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic diverticulosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dry heaves (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernia abdominal wall (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0)
Edema extremities (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 8 (9) | 1 (1)
Injection site reaction (General disorders) | 20 (141) | 0 (0)
Weakness (General disorders) | 1 (2) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (2) | 0 (0)
Drug allergy (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Oral thrush (Infections and infestations) | 1 (1) | 0 (0)
Otitis (Infections and infestations) | 1 (1) | 0 (0)
Pustules on hand (Infections and infestations) | 1 (1) | 0 (0)
Sinus infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (4) | 0 (0)
Upper respiratory tract infection viral NOS (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site tenderness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Abrasions (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bruise (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
LDH increased (Investigations) | 1 (1) | 0 (0)
Reticulocyte count increased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Groin discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leg cramps (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Swollen ankles (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Numbness (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Taste alteration (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral burning on micturition (Renal and urinary disorders) | 1 (1) | 0 (0)
Urination pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Spotting vaginal (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Congestion pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythematous rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Facial flushing (Vascular disorders) | 1 (2) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT01309230/Prot_SAP_000.pdf